CLINICAL TRIAL: NCT05860569
Title: A Multi-center, Open Label, Multi-arm, Dose Ascending Clinical Trial for Evaluation of Safety and Tolerance of Gene Therapy Drug GC304 in the Treatment of Primary Hypertriglyceridemia Patients With History of Acute Pancreatitis
Brief Title: Safety Evaluation of Gene Therapy Drug in the Treatment of Primary Hypertriglyceridemic Patients With Recurrent Pancreatitis
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: GeneCradle Inc (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: JL-GC304-01
Record Dates: First submitted 2023-04-23; First posted 2023-05-16 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-07

CONDITIONS: Hypertriglyceridemia, Familial
MeSH Terms: conditions — Hyperlipoproteinemia Type IV

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Cohort 1 (Experimental): 3.0x10^12 vg/kg of GC304 delivered one-time intravenously (n=3)
  Interventions: Genetic: GC304
- Cohort 2 (Experimental): 1.0x10^13 vg/ kg of GC304 delivered one-time i intravenously (n=3)
  Interventions: Genetic: GC304
- Cohort 3 (Experimental): 3.0x10^13 vg/ kg of GC304 delivered one-time i intravenously (n=3)
  Interventions: Genetic: GC304

INTERVENTIONS:
Genetic: GC304 — Self-complementary adeno-associated virus serotype 5 (AAV5) carrying a codon-optimized LPL coding sequence(coLPL) driven by a liver-specific promoter (LP)

SUMMARY:
The study will evaluate safety and tolerance of intravenous delivery of GC304 gene therapy drug as a treatment of primary hypertriglyceridemic patients with previous onset of acute pancreatitis.

DETAILED DESCRIPTION:
The purpose of this trial is to evaluate safety and tolerance of gene therapy drug GC304 in primary hypertriglyceridemic patients who have loss of function mutations in GPIHBP1 or LPL genes, with previous onset of acute pancreatitis.

Open-label, dose-escalation clinical trial of GC304 will be conducted in China. GC304 will be administrated intravenously. Short-term safety will be evaluated in 52 weeks and enter long-term follow-up study of 5 years at will. Patients will be tested at baseline and followed up on various time points.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed as primary hypertriglyceridemia poorly managed by regular treatment and dietary control, with episode of acute pancreatitis twice or once of severe acute pancreatitis within 5 years;
* Fasting plasma triglycerides (TG) levels above 5.65 mmol/L (intake of dietary fat <30 g within 24 hours before blood taken);
* Homozygous or heterozygous mutations in GPIHBP1 or LPL genes by genetic screening;
* The patients within reproductive age take effective contraceptive measures voluntarily entering screening stage until 6 months after the trial;
* The patients fully understand and are able to comply with the requirements of the treatment and are willing to complete the trial as planned, including voluntary compliance with the trial procedures, acceptance of low-fat dietary requirements, and provide of biological samples.
* Be able to understand the procedures and methods of the trial and voluntarily participate with the signature of the informed consent by the patient or his/her guardian.

Exclusion Criteria:

* Patient who is known to be allergic to any ingredient of a trial drug (including immunosuppressants) or has any disease prohibited from the treatment;
* Patient who is having active bacteria, fungi, viruses or other infections;
* Patient who is intolerant of immunosuppressive drugs or steroids;
* Patient who is with any of the following clinical history of serious illness or existing serious illness:

  1. unrelieved abdominal pain caused by acute onset of pancreatitis or by other causes；
  2. disease history of malignancy or currently suffering from any malignant tumor;
  3. autoimmune diseases;
  4. disease history of epilepsy or mental illness (e.g. schizophrenia, depression, mania, anxiety, etc.);
  5. heart diseases: cardiomyopathy and myocarditis; structural heart diseases; coronary heart disease (acute coronary syndrome, myocardial infarction); pericardial disease; severe arrhythmias (severe tachycardia requiring pacemakers, severe rapid arrhythmias, and other arrhythmias beyond the control of medications) ; New York Heart Association (NYHA) classification heart function grading ≥III or Left Ventricular Ejection Fraction (LVEF) ≤50%;
  6. poorly controlled diabetes (fasting blood glucose ≥11.1mmol/L);
  7. with systolic blood pressure (SBP) > 150mmHg and/or diastolic blood pressure (DBP) > 100mmHg after treatment with a stable dose (at least 4 weeks) of antihypertensive drugs;
* The results of the laboratory examination at screening meet either of the following:

  1. Aspartate transaminase (AST) or alanine transaminase (ALT) > 2 × upper limit of normals (ULN);
  2. Total bilirubin > upper limit of normals (ULN);
  3. Creatinine > upper limit of normals (ULN);
  4. Phosphatase kinase > 2 × upper limit of normals (ULN);
  5. Glomerular filtration rate estimate < 50 mL/min (estimated by the Cockroft-Gault formula);
  6. Positive hepatitis B surface antigen, positive hepatitis C antibody, positive HIV antibody or positive syphilis spiral antibody before or during screening;
  7. A positive blood pregnancy test;
* AAV5 neutralizing antibody levels above 1:100
* Person who has used a clinical trial drug within 1 month (30 days) prior to screening, or who plans to participate in other clinical trials during the trial period;
* Blood loss/donation of more than 400 mL (except for female physiological blood loss) within 3 months (90 days) before screening, and receiving blood transfusion or using blood products;
* Person who has undergone major surgery within 3 months (90 days) prior to screening, or who has undergone surgery that could significantly affect the course or safety evaluation of the trial drug;
* Alcohol consumption was high in the first 3 months (90 days), i.e. the average alcohol intake was greater than 3 units/day (Male) or 2 units/days (female) (1 unit = 18ml alcohol, such as beer 360 ml with 5% alcohol, 12% wine 150ml, 40% liquor 45ml); or who cannot abstain from drinking during the trial;
* Women who are pregnant, pregnant or breastfeeding, or all persons of reproductive age who are unable to take effective contraceptives until 3 months after the completion of the study;
* Patients who have poor compliance or who may not be able to complete the test for other reasons, or whom the investigator considers inappropriate to participate in the trial.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 7 (Estimated)
Dates: Start 2024-09-20 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability]) | 12 weeks
  Frequency of treatment-related adverse events (AEs), serious adverse events (SAEs), and changes from baseline in relevant clinical laboratory tests
The incidence of dose limited tolerance (DLT) | 12 weeks

SECONDARY OUTCOMES:
Changes of plasma triglyceride levels from baseline | 12 weeks
The proportion of patients who stop using lipid-lowering medications; | 12 weeks
Copy numbers of viral vector DNA [Shedding of viral vectors]; | 12 weeks
Titers of antibody against viral vector | 12 weeks
Titers of antibody against LPL (lipoprotein lipase) protein | 12 weeks

OTHER OUTCOMES:
Changes of LPL activity in post-heparin plasma from baseline; | 52 weeks
Frequency of onset of acute pancreatitis after administration of GC304; | 52 weeks
Changes of plasma triglyceride levels from baseline； | 52 weeks
The proportion of patients who stop taking hypolipidemic drugs; | 52 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Union Medical College, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No